CLINICAL TRIAL: NCT03926208
Title: Randomized Trial of Dilute Betadine Soak and Scrub for Foot and Ankle Surgery
Brief Title: Dilute Betadine Soak and Scrub for Foot and Ankle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Kamran S Hamid, MD, Principle Investigator, M.D. MPH, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18021801-IRB02
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Infection; Postoperative Complications
Keywords: Betadine; Foot; Ankle; Nail fold; Scrub; Infection; Prevention; Postoperative
MeSH Terms: conditions — Postoperative Complications; Infections

STUDY DESIGN:
Intervention Model Description: One group will be randomized to receive a betadine soak and scrub (in addition to the standard of care) prior to surgery. The control group will receive the standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Subjects in this group will receive the standard chlorhexadine prep of the foot (standard of care) prior to surgery, and a cotton swab will be collected from the hallux nail fold.
  Interventions: Procedure: Clorhexadine scrub
- Soak and Scrub (Experimental): In addition to the standard chlorhexadine prep of the foot prior to surgery, subjects in this group will also receive a betadine soak and scrub of the foot, and a cotton swab will be collected from the hallux nail fold.
  Interventions: Procedure: Soak and Scrub

INTERVENTIONS:
Procedure: Soak and Scrub — Betadine soak and scrub in addition to standard clorhexadine scrub (standard of care).
  Arms: Soak and Scrub
Procedure: Clorhexadine scrub — Clorhexadine scrub (standard of care).
  Arms: Control

SUMMARY:
Infection and wound complications are the most common complications following orthopaedic foot and ankle procedures, and the infection rate following these procedures is higher than in procedures involving other areas of the body.The purpose of this randomized controlled trial is to determine whether a standard chlorhexidine prep can be augmented with a soak & scrub of the foot in dilute betadine to reduce the rate of positive cultures from the hallux nail fold prior to surgery.

DETAILED DESCRIPTION:
Infection and wound complications are the most common complications following orthopaedic foot and ankle procedures, and the infection rate following these procedures is higher than in procedures involving other areas of the body. This is at least in part because the anatomy of the human foot presents inherent challenges for preoperative sterilization techniques due to the many folds and crevices associated with the toes. In particular, the nail folds of the toes are known to harbor large amounts of bacteria.

A systematic review and meta-analysis of previous studies that have investigated the efficacy of various foot and ankle preparation agents (including alcohol, chlorhexidine, chloroxylenol, and iodine/iodophors) showed that no single agent or combination of agents eliminates positive culture growth to undetectable levels for all patients. Articles have suggested superiority of a chlorhexidine prep solution over other types of preps; hence, chlorhexidine prep is now considered the gold standard at many institutions. But even a chlorhexidine prepped foot has been shown to contain culturable bacteria in the nail folds in 30% of cases.

The purpose of this randomized controlled trial is to determine whether a standard chlorhexidine prep can be augmented with a soak & scrub in dilute betadine to reduce the rate of positive cultures from the hallux nail fold.

It is hypothesized that in comparison to feet receiving the standard chlorhexadine prep, feet receiving the standard prep plus the betadine soak & scrub will be less likely to have culture positive swabs of the hallux nail fold.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Patient requires a foot or ankle operative procedure
3. Patient provides informed consent

Exclusion Criteria:

1. Patient refuses
2. Patient is incarcerated, incapacitated, or otherwise unable to provide appropriate informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamran S Hamid, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers.

REFERENCES:
- [Background] Butterworth P, Gilheany MF, Tinley P. Postoperative infection rates in foot and ankle surgery: a clinical audit of Australian podiatric surgeons, January to December 2007. Aust Health Rev. 2010 May;34(2):180-5. doi: 10.1071/AH08687. PMID 20497730
- [Background] Donley BG, Philbin T, Tomford JW, Sferra JJ. Foot and ankle infections after surgery. Clin Orthop Relat Res. 2001 Oct;(391):162-70. doi: 10.1097/00003086-200110000-00017. PMID 11603664
- [Background] Physiology for Nursing Practice Physiology for Nursing Practice edited by Hinchcliff S Montague S Published by Bailliere Tindall 680pp pound9.95 0-7020-1194-0 [Formula: see text]. Nurs Stand. 1988 May 21;2(33):34. doi: 10.7748/ns.2.33.34.s62. PMID 27416219
- [Background] Hunter JG, Dawson LK, Soin SP, Baumhauer JF. Randomized, Prospective Study of the Order of Preoperative Preparation Solutions for Patients Undergoing Foot and Ankle Orthopedic Surgery. Foot Ankle Int. 2016 May;37(5):478-82. doi: 10.1177/1071100715623037. Epub 2015 Dec 17. PMID 26678427
- [Background] Ostrander RV, Botte MJ, Brage ME. Efficacy of surgical preparation solutions in foot and ankle surgery. J Bone Joint Surg Am. 2005 May;87(5):980-5. doi: 10.2106/JBJS.D.01977. PMID 15866959
- [Background] Sands K, Vineyard G, Platt R. Surgical site infections occurring after hospital discharge. J Infect Dis. 1996 Apr;173(4):963-70. doi: 10.1093/infdis/173.4.963. PMID 8603978
- [Background] Yammine K, Harvey A. Efficacy of preparation solutions and cleansing techniques on contamination of the skin in foot and ankle surgery: A systematic review and meta-analysis. Bone Joint J. 2013 Apr;95-B(4):498-503. doi: 10.1302/0301-620X.95B4.30893. PMID 23653955

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were enrolled until protocol requirements were met.
Groups:
- Intervention: In addition to the standard chlorhexadine prep of the foot prior to surgery, subjects in this group will also receive a betadine soak and scrub of the foot, and a cotton swab will be collected from the hallux nail fold.
  Soak and Scrub: Betadine soak and scrub in addition to standard clorhexadine scrub (standard of care).
Period: Overall Study
Arm/Group | Control | Intervention
Started | 119 | 123
Completed | 119 | 123
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 119 | 123 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (16.5) | 51.2 (16.5) | 49.5 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 69 | 135
  Male | 53 | 54 | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 119 | 123 | 242
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 29.2 (6.8) | 29.3 (7.1) | 29.2 (7.0)
Splint [Count of Participants; unit: Participants] | 28 | 27 | 55

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Culture Growth
Description: Cotton swab of hallux nail fold. Culture of any microorganisms found. The results indicate the number of patients with positive bacterial culture growth.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 119 | 123
Participants | 32 | 33

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the patients global period (3 months) from the surgery date.
Description: Adverse events were monitored at every clinic visit after surgery.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/123
Other Adverse Events (participants affected / at risk) | 8/119 | 9/123
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=119) | Intervention (N=123)
Deep SSI (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) — Deep SSI was defined as similar symptoms treated with incision and debridement in the operating room.
Superficial Surgical Site Infection (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9) — Superficial surgical site infections or wound at risk was defined as peri-incisional erythema, redness, dehiscence, and/or drainage that was managed with oral antibiotics on an outpatient basis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03926208/Prot_SAP_ICF_000.pdf